CLINICAL TRIAL: NCT00277511
Title: Prospective, Multinational, Multicenter, Non-Comparative, Open Study With a 6 Months Follow-up Period to Demonstrate the Efficacy and Safety of Oral Levofloxacin 500 mg Once Daily in the Treatment of Chronic Bacterial Prostatitis (CBP)
Brief Title: Levofloxacin, Chronic Bacterial Prostatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR355/3036
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Prostatitis
MeSH Terms: conditions — Prostatitis | interventions — Levofloxacin

INTERVENTIONS:
Drug: Levofloxacin

SUMMARY:
Primary objective:

* To investigate the microbiological efficacy, assessed as eradication rate based on microbiologically evaluable patients 1 month post treatment with oral Levofloxacin 500 mg in male adults with chronic bacterial prostatitis (CBP, category II)

Secondary objectives:

* To investigate the microbiological efficacy, assessed as eradication rate based on microbiologically evaluable patients 6 months post treatment with oral Levofloxacin 500 mg in male adults with chronic bacterial prostatitis (CBP, category II).
* To assess the clinical response rate based on resolution of signs and symptoms after 2 weeks of treatment; 5-12 days, 1 month, 3 months and 6 months post treatment with oral Levofloxacin 500 mg in male adults with chronic bacterial prostatitis (CBP, category II).
* To assess the safety of Levofloxacin 500 mg on the basis of adverse events, standard clinical chemistry, hematology, urinalysis and vital signs in male adults with chronic bacterial prostatitis (CBP, category II).

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for enrollment into the study:

* A clinical diagnosis of chronic prostatitis as evidenced by the following criteria:

  * clinical signs and symptoms of prostatitis and
  * a history of chronic prostatitis as defined as: symptomatic prostatitis (a clinical diagnosis of prostatitis having been made for at least one previous episode which episode having lasted four weeks or two or more other episodes during the previous twelve months) and leucocyturia greater/equal 10 WBC/HPF x 400
* Laboratory evidence of prostatitis
* Candidate is appropriate for oral therapy.
* OTC medications for chronic prostatitis (other than antibiotics), which the subject has been receiving must continue throughout the study at the same dose or be discontinued prior to study entry.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Need for parenteral therapy for the treatment of chronic bacterial prostatitis (CBP, Category II)
* Subjects with pathogen known or suspected to be resistant to the study drug
* Requirement for a second systemic antibacterial regimen
* Any condition which may interfere with the evaluation of the study drug including transurethral prostatectomy within 6 months of enrollment, the presence of a permanent transurethral catheter or a history of cystostomy or nephrostomy
* Taking medication that may effect bladder or prostate function (e.g. hormone therapy anticholinergics or alpha-blocker)
* Patients not receiving saw palmetto at the time of study entry should not start treatment with saw palmetto within 10 weeks of study entry
* Known prostatic carcinoma
* The presence of another infection requiring therapy with an antibacterial other than the study drug
* Greater than 24 hours of potentially effective therapy within seven days prior to study when there is documented evidence of a resistant organism or clinical failure after five or more days of previous antibacterial therapy
* History of hypersensitivity to the investigational product or to drugs with similar chemical structures
* History of tendonitis or tendon rupture
* Treatment with other quinolones in the last 14 days before study entry
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Treatment with any investigational product in the last 30 days before study entry
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* History of drug or alcohol abuse
* Impaired hepatic function, as shown by:

  * AST (SGOT) greater/equal 3 times the upper limit of the reference range
  * ALT (SGPT) greater/equal 3 times the upper limit of the reference range
  * bilirubin greater 51 µmol/l, i.e., greater 3 mg/dl (except of Gilbert disease)
  * hepatic encephalopathy
* Impaired renal function, as shown by either creatinine clearance smaller 50 ml/min or undergoing hemodialysis or peritoneal dialysis (creatinine clearance may be estimated by formula or nomogram)
* Underweight (40 kg or less)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-03

PRIMARY OUTCOMES:
Primary efficacy data will be determined by eradication rate based on microbiologically evaluable subjects, evaluated for each pathogen and subject. | determined at 1 month follow-up

SECONDARY OUTCOMES:
Secondary efficacy data will be determined by microbiological eradication rate | at 6 months follow-up
clinical response rate based on resolution of signs and symptoms | after 2 weeks of treatment and during follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Roscher, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Berlin, Germany